CLINICAL TRIAL: NCT03027167
Title: Outcomes Study to Determine the Incidence of Symptomatic DVT/PE in Patients Receiving Aspirin With Mechanical Compression Devices Versus Aspirin Alone Following Knee and Hip Arthroplasty
Brief Title: Outcomes Study in Patients Receiving Aspirin With Mechanical Compression Devices Versus Aspirin Alone Following Knee and Hip Arthroplasty
Acronym: PDAS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Medical Compression Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201608075
Record Dates: First submitted 2017-01-03; First posted 2017-01-23 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: DVT - Deep Vein Thrombosis; PE - Pulmonary Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin and MCDs (Active Comparator): ASA with MCDs- Patients will receive MCDs intraoperatively and during the immediate post-operative recovery period, and will receive MCDs for a period of 10 days post-surgery. ASA 325mg BID will be prescribed for a period of 6 weeks.
  Interventions: Drug: Aspirin; Device: (Post- discharge) Mechanical Compression Device
- Aspirin only (Experimental): ASA only- Patients will receive MCDs intraoperatively and during the immediate post-operative recovery period, and will NOT receive MCDs after being discharged from hospital. ASA 325mg BID will be prescribed for a period of 6 weeks.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin
Device: (Post- discharge) Mechanical Compression Device
  Other Names: MCD, compression pump, mobile pumps
  Arms: Aspirin and MCDs

SUMMARY:
The Purpose is to compare the safety and efficacy of the use of aspirin(ASA) with medical compression devices versus aspirin alone for venous thromboprophylaxis following knee and hip arthroplasty.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE), which includes deep vein thrombosis (DVT) and pulmonary embolism (PE), is the most common complication occurring in association with knee and hip arthroplasty procedures due to an activation of the clotting cascade during bone and intramedullary canal preparation.DVT rates ranging from 4% to 15 % and PE rates ranging from 0.83% to 3% have been reported, with fatal PE rates reduced with the use of postoperative anticoagulation. The high risk of thromboembolic disease has led to recommendations that pharmacoprophylaxis be considered routinely. • The combination of short duration outpatient anticoagulation, early mobilization, and mechanical prophylaxis has recently been studied at our institution (Barnes-Jewish Hospital) and has been effective in prophylaxis against VTE. Current American College of Chest Physician (ACCP) guidelines recommend that a longer duration of outpatient anticoagulation following TKA / THA surgery may further reduce the risk of VTE.

Shorter patient hospitalizations and earlier discharge require an outpatient VTE prophylaxis regimen that is simple, effective, easy to monitor, predictable, and has a high patient compliance. Currently, "routine" risk patients receive a combination of ASA 325mg BID (twice daily) for a period of 6 weeks, and portable, mobile pneumatic compression devices (MCDs) for a period of 10 days post- surgery.The study is testing to see whether the use of ASA alone can be equally effective versus the use of ASA with MCDs in "routine" risk patients following total joint arthroplasty.Patients are enrolled fpr 6 months following surgery, and data collection occurs pre-surgery, 14 days after surgery, at the 4-8 wk visit and finally, at 6 months post surgery. We are evaluating the stated outcomes over this 6 month period.

ELIGIBILITY:
Inclusion Criteria:

* All total knee arthroplasty (TKA), unicompartmental knee arthroplasty (UKA), total hip arthroplasty (THA), and surface replacement arthroplasty (SRA) patients age 18 or older and undergoing an elective primary or revision procedure will be eligible to participate in this study.

Exclusion Criteria:

Patients will be excluded if they are on chronic Coumadin therapy, require prolonged immobilization (i.e. cast/knee immobilizer; inability to be full weight-bearing and out of bed on postoperative day 1), and are scheduled to have multiple surgeries in close proximity to one another. Based on our institution's risk stratification protocol, all patients deemed "high risk" and meeting one of the following criteria will also be excluded as they would receive Coumadin for VTE prophylaxis:

1. Patients will be excluded if they are on chronic Coumadin therapy
2. History of DVT/PE
3. Active Cancer
4. Hypercoaguable States (Protein C, Protein S, Factor V Leiden, etc.)
5. Family history of thrombosis -note: we may remove this criteria after further discussion
6. Patients requiring prolonged immobilization (i.e. cast/knee immobilizer),
7. Patients having multiple surgeries in close proximity to one another.
8. Patients with known allergy or hypersensitivity to Aspirin or Platelet count < 60, 000
9. Patients receiving bilateral joint replacement

Patients who consent to the study and cancel/do not have a surgery scheduled within six months of signing the consent form will not be included. immobilization (i.e. cast/knee immobilizer; inability to be full weight-bearing and out of bed on postoperative day 1), and are scheduled to have multiple surgeries in close proximity to one another. Based on our institution's risk stratification protocol, all patients deemed "high risk" and meeting one of the following criteria will also be excluded as they would receive Coumadin for VTE prophylaxis:

1. Patients will be excluded if they are on chronic Coumadin therapy
2. History of DVT/PE
3. Active Cancer
4. Hypercoaguable States (Protein C, Protein S, Factor V Leiden, etc.)
5. Family history of thrombosis -note: we may remove this criteria after further discussion
6. Patients requiring prolonged immobilization (i.e. cast/knee immobilizer),
7. Patients having multiple surgeries in close proximity to one another.
8. Patients with known allergy or hypersensitivity to Aspirin or Platelet count < 60, 000
9. Patients receiving bilateral joint replacement

Patients who consent to the study and cancel/do not have a surgery scheduled within six months of signing the consent form will not be included. (Note: The surgery does not have to occur within six months of signing the consent form but must be scheduled/re-scheduled within six months of signing the consent form.) If these patients decide to schedule surgery after the six months has passed, they will be re-consented at the time they schedule surgery.

Patients who are not willing to participate will also be excluded from the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
VTE/PE | 6 months
  Using the MCS (Mobile Compression Systems) Mobile Pumps system for 10 days after surgery from hospital combined with 6 weeks of aspirin will prove superior to the use of 6 weeks of aspirin in the prophylaxis of VTE/PE in standard risk joint arthroplasty patients. Efficacy will be measured in relation to previously published clinical trials with these agents and with previous patient cohorts at our institution.

SECONDARY OUTCOMES:
Cessation of anticoagulation therapy for any reason | 6 months
  Patient reported data will be collected to capture this information.
Readmission to the hospital for any VTE event or surgical site complication in relation to VTE prophylaxis therapy | 6 months
  Electronic Medical Records will be reviewed and patient reported data will be collected

IPD SHARING:
Plan to Share IPD: Undecided